CLINICAL TRIAL: NCT02694198
Title: Fetal Fibronectin as a Predictor of Successful Induction of Mid-trimester Abortion
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Amr Ahmed Mahmoud Riad, Lecturer of obstetrics and gynecology, Ain Shams Maternity Hospital
Other Study IDs: fetal fibronectin
Record Dates: First submitted 2016-02-24; First posted 2016-02-29 (Estimated); Results first posted 2016-04-06 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Medical; Abortion, Fetus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: fetal fibronectin measurement — All patients will be put in the dorsal lithotomy position.Using a proper light source and sterile gloves, a sterile speculum free of lubricants will be placed into the vagina before vaginal examination by senior resident and the special Dacron swab from the FFN kit will be used to collect a sample of secretions from the posterior fornix. The sample should be obtained prior to collection of any vaginal wet preparations, before any cervical manipulation or cervical cultures, and if enough amount of fluid (about 2 ml) is not found, vagina will be washed with 2 ml of normal saline.The swab will be placed in sterile plastic containers which will be stored until assayed quantitatively with an Enzyme-Linked Immuno Sorbant Assay.

SUMMARY:
Fetal Fibronectin as a Predictor of Successful Induction of Mid-trimester abortion.

DETAILED DESCRIPTION:
The population of the study will comprise 135 pregnant women attending Ain Shams University Maternity hospital at labor and delivery ward diagnosed with mid-trimester missed miscarriage confirmed by transabdominal ultrasound who will undergo termination by misoprostol.

Before entering the study, the purpose of this work will be clearly explained and verbal consent will be obtained from all patients enrolled in the study along with routine written informed consent as governed by the hospital rules.

All participants will be subjected to:

1. History taking:

   1. Personal history: age and special habits
   2. Obstetric history (parity, history of abortions, previous cerculage and preterm labor). Gestational Age will be assigned by means of a combination of menstrual dating and ultrasonographic evaluation.
   3. Past medical history (hypersensitivity to misoprostol, chronic adrenal insufficiency and inherited porphyrias).
   4. Past history of previous cesarean section or other operations as hysterotomy and myomectomy.
2. Examination:

   1. General examination: blood pressure, pulse, temperature, body weight.
   2. Abdominal examination: fundal level, presence of scar of previous operations, uterine contractions.
3. Investigations:

   1. Laboratory: complete blood count, c-reactive protein titre, blood group.
   2. Pelvic ultrasound: to assess fetal viability, amount of liquor, gestational age, position of the placenta.
4. Assessment of vaginal fetal fibronectin:

All Patients will be put in the dorsal lithotomy position.Using a proper light source and sterile gloves, a sterile speculum free of lubricants will be placed into the vagina before vaginal examination by senior resident and the special Dacron swab from the fetal fibronectin kit will be used to collect a sample of secretions from the posterior fornix. The sample will be obtained prior to collection of any vaginal wet preparations, before any cervical manipulation or cervical cultures, and if enough amount of fluid (about 2ml) is not found, vagina will be washed with 2ml of normal saline.The swab will be placed in sterile plastic containers which will be stored until assayed quantitatively with an Enzyme-Linked Immuno Sorbant Assay.

According to Ain Shams University Maternity Hospital protocol, termination of pregnancy will be conducted as an inpatient procedure. Termination of pregnancy will be performed using misoprostol tablets (Misotac® Sigma 200 mcg per tablet). Misoprostol tablets will be introduced by vaginal routes initially (total 800 mcg). Following the initial dose, 2 misoprostol tablets (400 mcg) will be inserted into the vagina every 4 hours to a maximum of four doses. If the woman does not have adequate contractions, within 8 hours following the last dose, the same regimen will be repeated over the following 24 hours without the loading dose.

The induction to expulsion period will be defined as the time from commencement of misoprostol until fetal expulsion without exerting any fetal traction by caregiver. After expulsion of the fetus, the patients will receive 30 units of oxytocin on 500 cc Ringer solution slowly by intravenous infusion over 30 minutes for expulsion of the placenta. Surgical evacuation will be done when indicated.

The kits used to measure level of fetal fibronectin in vaginal sample (ZYMUTEST Fibronectin kits) were provided from Hyphen BioMed corporation , France. The ZYMUTEST Fibronectin kit is an one-step enzyme immuno-assay for measuring human Fibronectin in plasma, or in any fluid where fibronectin can be present.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy.
* 14-24 weeks gestation..
* Missed miscarriage

Exclusion Criteria:

* History of pulmonary, hepatic, renal, or cardiovascular diseases.
* History of previous cesarean section and other uterine surgeries as hysterotomy and myomectomy.
* Inevitable abortion.
* Placenta covering internal os.
* History of any cervical surgery as cervical amputation, cauterization or dilatation.
* Premature rupture of membranes.
* Any vaginal bleeding.
* Contraindications for misoprostol as hypersensitivity to misoprostol, chronic adrenal insufficiency and inherited porphyrias.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 135 pregnant women attending Ain Shams University Maternity hospital at labor and delivery ward diagnosed with mid-trimester missed miscarriage confirmed by transabdominal ultrasound who will undergo termination by misoprostol
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Mid-trimester Abortion: The population of the study comprised 135 pregnant women attending Ain Shams University Maternity hospital at labor and delivery ward diagnosed with mid-trimester missed miscarriage confirmed by transabdominal ultrasound who will undergo termination by misoprostol
Period: Overall Study
Arm/Group | Mid-trimester Abortion
Started | 135
Completed | 135
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Depending on Francesco et al., 2005 who found that Fetal fibronectin positive test in 19 among 270 (7.0%) in women undergoing mid-trimester abortion. Assuming α=0.05 and confidence interval (CI)= 10.0% and by using PASS 11th release the minimal sample size is 120. With a possible 10.0% drop out of cases, the enrolled cases would be 135 cases.
Arm/Group | Mid-trimester Abortion
Number analyzed (Participants) | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.4 (4.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135
  Male | 0
Body mass index [Mean (Standard Deviation); unit: kilograms per squared meter] | 29.4 (2.31)
gestational age in weeks [Mean (Standard Deviation); unit: weeks] | 19.32 (1.91)
Outcome of induction of abortion [Number; unit: participants]
  abortion in less than 24 hours | 119
  abortion in more than 24 hours | 13
  failed induction | 3

OUTCOME MEASURES:

1. Primary Outcome: Cervicovaginal Fetal Fibronectin Level
Description: mean cervicovaginal fetal fibronectin level in women undergoing midtrimesteric induction of abortion
Time Frame: 72 hours
Population: Depending on Francesco et al., 2005 who found that Fetal fibronectin test positive in 19 among 270 (7.0%) women undergoing mid-trimester abortion. Assuming α=0.05 and confidence interval (CI)= 10.0% and by using PASS 11th release the minimal sample size is 120. With a possible 10% drop out of cases, the enrolled cases would be 135 cases.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Mid-trimester Abortion
Number analyzed (Participants) | 135
nanogram per milliliter | 39.4 (7.9)

2. Primary Outcome: Relation of Cervicovaginal Fetal Fibronectin Level to Duration of Induction of Abortion
Description: Difference between women who expulsed the fetus within 24 hours and women who expulsed the fetus in more than 24 hours as regarding cervicovaginal fetal fibronectin level (ng/ml)
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Mid-trimester Abortion
Number analyzed (Participants) | 135
nanogram per milliliter
  women aborted within 24 hours n=129 | 39.3 (7.71)
  women aborted in more than 24 hours or failed n=6 | 40.4 (11.2)

ADVERSE EVENTS:
Time Frame: All participants were closely monitored during the process of induction of abortion and over the following 24 hours following spontaneous expulsion or surgical removal of the placenta.
Arm/Group | Mid-trimester Abortion
Serious Adverse Events (participants affected / at risk) | 0/135
Other Adverse Events (participants affected / at risk) | 118/135
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mid-trimester Abortion (N=135)
Need for surgical removal of placenta (Surgical and medical procedures) | 87 (87)
Shivering (General disorders) | 5 (5)
Fever (General disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 12 (12)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No